CLINICAL TRIAL: NCT00669032
Title: Random, Phase IV, Multicentre, Double Blind, Placebo Controlled, Parallel Study to Assess Long-term Efficacy and Safety of Repeated Intraarticular Injections of Hyaluronic Acid (ADANT®) in Patients With Knee OA of the Knee
Brief Title: Efficacy and Safety of Repeated Intraarticular Injections of Hyaluronic Acid in Patients With OA of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tedec-Meiji Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TM-ME3710/304; 2006-001854-28 (EudraCT Number)
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- hyaluronic acid (Experimental): Cycles of 5 injections of hyaluronic acid at specified intervals
  Interventions: Device: Hyaluronic acid
- Placebo (Placebo Comparator): Cycles of 5 injections of saline at specified intervals
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Hyaluronic acid — 3 cycles of 5 hyaluronic acid injections, with a 6 month interval between each one. A 4th treatment cycle of five injections will be carried out at the end of one year
  Arms: hyaluronic acid
Other: Placebo — 3 cycles of 5 saline solution injections, with a 6 month interval between each one. A 4th treatment cycle of five injections will be carried out at the end of one year
  Arms: Placebo

SUMMARY:
The main objective is the long-term comparison (3 years and 4 months) of the efficacy and safety of repeated intra-articular administration of hyaluronic acid in the treatment of osteoarthritis of the knee.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of repeated injections of hyaluronic acid compared with placebo over a period of 40 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 45 years of age
* Out-patient diagnosed with primary osteoarthritis of the femorotibial medial joint of the knee with clinical and radiological (Kellgren grade II-III) ACR diagnosis
* Joint Space Width (JSW) > 2mm
* Overall pain greater or equal to 55mm (VAS - Visual Analogue Scale 100mm) recorded in the knee,by the patient at any time during the week prior to the evaluation

Exclusion Criteria:

* Overweight patients (body mass index > 32).
* Pregnant and lactating women. Women of child-bearinge age not using effective contraception
* Patients who have received intra-articular hyaluronic acid within the previous year and/or intra-articular steroids or articular lavage in the chosen knee,within the previous 3 months prior to their inclusion in the study.
* AINE administration within the 14 days prior to their inclusion in the study.
* Administration of glucosamine sulphate, chondroitin sulphate and diacerein within the 3 months prior to their inclusion in the study.
* Immunocompromised patients or patients receiving systemic immunosuppressive therapy.
* Patients with known sensitivity to HA, parcetamol or AINEs permitted as rescue medication.
* Patients who have received any investigational drug within 30 days prior to visit 1, or who are scheduled for the administration of an investigational drug other than the protocol product during this study.
* Patients with severely impaired central nervous system.
* Patients with coagulation alterations, despite receiving treatment.
* Patients with secondary osteoarthritis of the knee
* Patients having previously received surgery, including arthroscopy
* Patients with articular inflammatory disease

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2003-10; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Navarro Sarabia, Principal Investigator

REFERENCES:
- [Result] Navarro-Sarabia F, Coronel P, Collantes E, Navarro FJ, de la Serna AR, Naranjo A, Gimeno M, Herrero-Beaumont G; AMELIA study group. A 40-month multicentre, randomised placebo-controlled study to assess the efficacy and carry-over effect of repeated intra-articular injections of hyaluronic acid in knee osteoarthritis: the AMELIA project. Ann Rheum Dis. 2011 Nov;70(11):1957-62. doi: 10.1136/ard.2011.152017. Epub 2011 Aug 17. PMID 21852252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting started in October 2003 and the last follow-up was performed on July 2009. This study enrolled patients from the Rheumatology Departments belonging to 19 centres located in Spain.
Pre-assignment Details: A total of 446 patients were screened, of whom 140 (31,4%) were screening failures. At the screening visit the patients were assessed by the blinded physician for fulfilment of the selection criteria, demographic characteristics and medical history. Knee radiographs were also obtained.
Groups:
- Hyaluronic Acid (Adant): Four cycles of 5 weekly intra-articular injections of 2.5ml 1% sodium hyaluronate with a follow-up of 6 months after the first and second cycles, and 1 year after the third and fourth cycles.
- Placebo: Four cycles of 5 weekly intra-articular injections of 2.5ml saline solution with a follow-up of 6 months after the first and second cycles, and 1 year after the third and fourth cycles.
Period: Overall Study
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Started | 153 | 153
Completed | 109 | 94
Not Completed | 44 | 59
Not completed — Lost to Follow-up | 6 | 5
Not completed — Lack of Efficacy | 8 | 19
Not completed — Withdrawal by Subject | 12 | 13
Not completed — Adverse Event | 12 | 16
Not completed — Physician Decision | 1 | 1
Not completed — No fulfilment of the selection criteria | 5 | 5

BASELINE CHARACTERISTICS:
Population: Considering a statistical power of 80% and assuming up to a 40% dropout rate, the sample size was planned to include a total of 300 patients (150 per treatment arm). Analysis was performed based on the modified intention-to-treat population. The imputation method for handling missing data was the last observation carried forward.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyaluronic Acid (Adant) | Placebo | Total
Number analyzed (Participants) | 153 | 153 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.2) | 63.9 (8.9) | 63.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 128 | 256
  Male | 25 | 25 | 50
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (2.7) | 28.7 (2.6) | 28.6 (2.7)
Duration knee osteoarthritis [Mean (Standard Deviation); unit: years] | 6.9 (6.8) | 8.1 (8.4) | 7.5 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Responders OARSI 2004 at the End of Follow-up
Description: Percentage of subjects with a clinical response according to Osteaorthritis Research Society International (OARSI) 2004 criteria at the end of follow-up. Patients were classified as responders if the pain or physical function scores decreased at least 50% and at least 20mm on the Visual Analogue Scale (VAS), or if two of the following three findings were recorded: a decrease in pain score of at least 20% or at least 10mm on the VAS, a decrease in physical function score of at least 20% and at least 10mm on the VAS, or an increase in the score of the patient's global assessment by at least 20% and at least 10mm on the VAS.
  The VAS is set between 0-100mm, higher values represent a worse outcome in all cases except for both patient and physician global assessments where higher values indicate a better outcome.
Time Frame: 40 months
Population: The modified intention-to-treat population included all randomly assigned patients with at least one efficacy assessment after randomisation.
Measure: Number; unit: percentage of responders
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of responders | 80.5 | 65.8
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.004, Chi-squared

2. Secondary Outcome: Responders OARSI 2004 at 7 Months Follow-up Visit
Description: Percentage of subjects with a clinical response according to Osteaorthritis Research Society International (OARSI) 2004 criteria at 7 months follow-up visit (6 months after first cycle). Patients were classified as responders if the pain or physical function scores decreased at least 50% and at least 20mm on the Visual Analogue Scale (VAS), or if two of the following three findings were recorded: a decrease in pain score of at least 20% or at least 10mm on the VAS, a decrease in physical function score of at least 20% and at least 10mm on the VAS, or an increase in the score of the patient's global assessment by at least 20% and at least 10mm on the VAS.
  The VAS is set between 0-100mm, higher values represent a worse outcome in all cases except for both patient and physician global assessments where higher values indicate a better outcome.
Time Frame: 7 months (6 months after first cycle)
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of responders | 71.1 | 67.8
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.525, Chi-squared

3. Secondary Outcome: Responders OARSI 2004 at 14 Months Follow-up Visit
Description: Percentage of subjects with a clinical response according to Osteaorthritis Research Society International (OARSI) 2004 criteria at 14 months follow-up visit (6 months after second cycle). Patients were classified as responders if the pain or physical function scores decreased at least 50% and at least 20mm on the Visual Analogue Scale (VAS), or if two of the following three findings were recorded: a decrease in pain score of at least 20% or at least 10mm on the VAS, a decrease in physical function score of at least 20% and at least 10mm on the VAS, or an increase in the score of the patient's global assessment by at least 20% and at least 10mm on the VAS.
  The VAS is set between 0-100mm, higher values represent a worse outcome in all cases except for both patient and physician global assessments where higher values indicate a better outcome.
Time Frame: 14 months (6 months after second cycle)
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of responders | 76.5 | 65.1
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.030, Chi-squared

4. Secondary Outcome: Responders OARSI 2004 at 21 Months Follow-up Visit
Description: Percentage of subjects with a clinical response according to Osteaorthritis Research Society International (OARSI) 2004 criteria at 21 months follow-up visit (6 months after third cycle). Patients were classified as responders if the pain or physical function scores decreased at least 50% and at least 20mm on the Visual Analogue Scale (VAS), or if two of the following three findings were recorded: a decrease in pain score of at least 20% or at least 10mm on the VAS, a decrease in physical function score of at least 20% and at least 10mm on the VAS, or an increase in the score of the patient's global assessment by at least 20% and at least 10mm on the VAS.
  The VAS is set between 0-100mm, higher values represent a worse outcome in all cases except for both patient and physician global assessments where higher values indicate a better outcome.
Time Frame: 21 months (6 months after third cycle)
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of responders | 77.9 | 67.8
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.049, Chi-squared

5. Secondary Outcome: Responders OARSI 2004 at 27 Months Follow-up Visit
Description: Percentage of subjects with a clinical response according to Osteaorthritis Research Society International (OARSI) 2004 criteria at 27 months follow-up visit (12 months after third cycle). Patients were classified as responders if the pain or physical function scores decreased at least 50% and at least 20mm on the Visual Analogue Scale (VAS), or if two of the following three findings were recorded: a decrease in pain score of at least 20% or at least 10mm on the VAS, a decrease in physical function score of at least 20% and at least 10mm on the VAS, or an increase in the score of the patient's global assessment by at least 20% and at least 10mm on the VAS.
  The VAS is set between 0-100mm, higher values represent a worse outcome in all cases except for both patient and physician global assessments where higher values indicate a better outcome.
Time Frame: 27 months (12 months after third cycle)
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of responders | 77.9 | 67.8
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.049, Chi-squared

6. Secondary Outcome: Responders OARSI 2004 at 34 Months Follow-up Visit
Description: Percentage of subjects with a clinical response according to Osteaorthritis Research Society International (OARSI) 2004 criteria at 34 months follow-up visit (6 months after fourth cycle). Patients were classified as responders if the pain or physical function scores decreased at least 50% and at least 20mm on the Visual Analogue Scale (VAS), or if two of the following three findings were recorded: a decrease in pain score of at least 20% or at least 10mm on the VAS, a decrease in physical function score of at least 20% and at least 10mm on the VAS, or an increase in the score of the patient's global assessment by at least 20% and at least 10mm on the VAS.
  The VAS is set between 0-100mm, higher values represent a worse outcome in all cases except for both patient and physician global assessments where higher values indicate a better outcome.
Time Frame: 34 months (6 months after fourth cycle)
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of responders | 81.2 | 65.1
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.002, Chi-squared

7. Secondary Outcome: Pain or Function Scores Reduction 50% (20mm) at the End of Follow-up
Description: Percentage of patients with a decrease in pain or physical function score of at least 50% and at least 20mm on the VAS at the end of follow-up.
  The VAS is set between 0-100mm, higher values represent a worse outcome.
Time Frame: 40 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of patients | 65.1 | 52.0
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.021, Chi-squared

8. Secondary Outcome: Overall Pain Reduction 20% (10mm) at the End of Follow-up
Description: Percentage of patients with a decrease in pain score of at least 20% or at least 10mm on the VAS at the end of follow-up.
  The VAS is set between 0-100mm, higher values represent a worse outcome.
Time Frame: 40 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of patients | 79.2 | 67.8
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.025, Chi-squared

9. Secondary Outcome: Function Improvement 20% (10mm) at the End of Follow-up
Description: Percentage of patients with a decrease in physical function score of at least 20% or at least 10mm on the VAS at the end of follow-up.
  The VAS is set between 0-100mm, higher values represent a worse outcome.
Time Frame: 40 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of patients | 70.5 | 57.9
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.023, Chi-squared

10. Secondary Outcome: Patient's Global Assessment Increase 20% (10mm) at the End of Follow-up
Description: Percentage of patients with an increase in the score of patient's global assessment by at least 20% and at least 10mm on the VAS at the end of follow-up.
  The VAS is set between 0-100mm, higher values represent a better outcome.
Time Frame: 40 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of patients | 74.5 | 57.9
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.002, Chi-squared

11. Secondary Outcome: Percentage of Patients Who Consumed Rescue Medication for Osteoarthritis
Description: Consumption of rescue medication (paracetamol/NSAID) for osteoarthritis throughout the study, an average of 40 months
Time Frame: Throughout the study, an average of 40 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
percentage of patients | 71.1 | 71.7
Statistical Analysis 1: Comparison: Hyaluronic Acid (Adant) vs Placebo; Test type: Superiority or Other; p = 0.9129, Chi-squared

12. Secondary Outcome: Mean Daily Dose of Paracetamol Consumption
Description: Mean daily dose of paracetamol consumption throughout the study, an average of 40 months
Time Frame: Throughout the study, an average of 40 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Number analyzed (Participants) | 149 | 152
mg/day | 408.8 (644.2) | 451.4 (925.8)

ADVERSE EVENTS:
Time Frame: 40 months
Description: Treatment safety and tolerability was evaluated based on the incidence and type of adverse events and the results of blood laboratory tests and physical examinations throughout the duration of the study. Safety analyses were performed in those patients who received at least one intra-articular injection (safety population).
Arm/Group | Hyaluronic Acid (Adant) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/153
Other Adverse Events (participants affected / at risk) | 11/153 | 11/153
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyaluronic Acid (Adant) (N=153) | Placebo (N=153)
Allergic reaction (Immune system disorders) | 3 (3) | 3 (3)
Pain at injection site (General disorders) | 6 (6) | 2 (2)
Bleeding at injection site (General disorders) | 2 (2) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Heaviness feeling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bleeding (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Control of rescue medication: patients were asked at every assessment visit about the frequency and doses of consumption, but it was not delivered in hand.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PIs is that the study results will be presented during scientific meetings or published in scientific journals with prior agreement with the sponsor.